CLINICAL TRIAL: NCT05918198
Title: Clinical Study of BCL-2 Inhibitor Venetoclax Combined With CAG in the Treatment of Refractory/Relapsed Acute Myeloid Leukemia
Brief Title: Clinical Study of Venetoclax Combined With CAG in the Treatment of Refractory/Relapsed Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Wen-Jing Yu, MD, Peking University People's Hospital, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDL2022-13
Record Dates: First submitted 2023-05-24; First posted 2023-06-26 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; CAG protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ven+CAG (Experimental): Venetoclax plus CAG regimen
  Interventions: Drug: Ven+CAG

INTERVENTIONS:
Drug: Ven+CAG — 100 mg on the first day, and then gradually increase to the target dose of 400 mg (100 mg d1, 200 mg d2, 400 mg d3) within 3 days; After that, the drug continued to be administered until the 14th day, 400 mg/day. When combined with CYP3A or P-gp inhibitors (mainly voriconazole in this study), adjust the venetoclax dose to 100 mg/day.
  Ara-C 10mg/m2, ih, q12h × 14d； Acla 20mg/d × 4d； G-CSF 5ug/kg × 14d (WBC > 30 × 10^9/L pause)
  Other Names: Venetoclax plus CAG regimen

SUMMARY:
The goal of this clinical trial is to test the safety and efficacy of venetoclax plus CAG regimen in refractory/relapsed acute myeloid leukemia patients.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

* Safety of Ven combined with CAG regimen in the treatment of relapsed/refractory AML patients
* Efficacy of Ven combined with CAG regimen in the treatment of relapsed/refractory AML patients Participants will receive therapy of venetoclax and CAG regimen (Ara-C, Acla and C C-GSF)

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age ≤ 75 years, male and female are not limited.
* According to bone marrow morphology and immunophenotype, it was diagnosed as acute myeloid leukemia ( WHO 2016 diagnostic criteria).
* Morphological recurrence after complete remission (CR) (leukemic cells in the peripheral blood of CR patients or more than 5% of the blasts in the bone marrow or new pathological hematopoiesis or extramedullary leukemic cell infiltration) or acute myeloid leukemia patients who did not achieved CR after 1 cycle of chemotherapy.
* The ECOG (Eastern Cancer Cooperation Group of the United States) PS score is 0-1.
* The expected survival time is ≥ 12 weeks.
* Female patients of childbearing age need to undergo pregnancy examination before receiving chemotherapy, and must agree to take effective contraceptive measures during treatment.
* Subjects volunteered to participate, fully informed consent, signed an informed consent, and good compliance.

Exclusion Criteria:

* Other malignant hematological diseases that do not conform to the diagnosis of acute myeloid leukemia.
* Allergy to any drugs involved in the project.
* History of serious cardiovascular and cerebrovascular diseases: ① Congestive heart failure, unstable angina pectoris, myocardial infarction, stroke or poorly controlled arrhythmia with NYHA grade II or above occurred within 12 months before enrollment，LVEF (left ventricular ejection fraction)<50% by color Doppler ultrasound，Corrected QT interval (QTc)>480ms (calculated by Fridericia method, if the QTc is abnormal, it can be detected continuously for 3 times every 2 minutes, and the average value is taken)，Hypertension difficult to control by drugs (systolic blood pressure (BP) ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg) (based on the average of ≥ 3 BP readings obtained from ≥ 2 measurements)，Have had hypertensive crisis or hypertensive encephalopathy in the past.
* There are other obvious bleeding tendencies or evidence of major coagulation disorders: ①Hemoptysis of any reason occurred within 2 weeks before enrollment，② Thrombosis or embolism occurred within 6 months before enrollment，③ Anticoagulant therapy for therapeutic purposes (except low molecular weight heparin therapy) be used within 2 weeks before enrollment④ Antiplatelet therapy is required.
* Abnormal liver function: total bilirubin>3 mg/dL；Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 5 × Upper limit of normal value (ULN).
* Abnormal renal function: serum creatinine ≥ 1.5 × ULN, or the creatinine clearance rate (CrCl) calculated according to Cockroft-Gault formula is less than 60 mL/min (if the calculated CrCl is less than 60 mL/min, the researcher may ask to confirm the 24-hour CrCl, in this case, the subjects with 24-hour CrCl less than 60 mL/min should be excluded).
* Other serious diseases that may limit the patient's participation in this clinical trial (including but not limited to other malignant tumors, active infection, serious uncured wounds, active ulcers and untreated fractures, history of human immunodeficiency virus infection, and receiving allogeneic stem cells or solid organ transplantation).
* Cannot swallow pills, malabsorption syndrome or any condition that affects gastrointestinal absorption.
* Other clinical trials are being conducted.
* Unable to understand or cooperate to complete the research protocol.
* Pregnant and lactating patients
* Other situations that the researcher believes are not suitable for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
CR/CRi rate | 2 to 3 weeks after the end of cycle 1 (each cycle is 14 days)
  the rate of complete remission or complete remission with incomplete hematologic recovery
CR/CRi rate | 2 to 3 weeks after the end of cycle 2 (each cycle is 14 days)
  the rate of complete remission or complete remission with incomplete hematologic recovery

SECONDARY OUTCOMES:
MRD status | 2 to 3 weeks after the end of cycle 1 (each cycle is 14 days)
  MRD-positive status was defined as FCM positivity in two consecutive BM samples at a 2-week interval, PCR positivity in two consecutive BM samples at a 2-week interval, or both FCM and PCR positivity in a single BM sample after the first-month post-HSCT. Positive FCM was defined as >0.01% of cells with a LAIPs phenotype in >1 BM samples after transplantation. The expressions of leukemia-associated genes were evaluated by TaqMan-based RT-PCR, including Wilms' tumor gene 1 (WT1) and genes which were determined in the diagnostic specimens.
MRD status | 2 to 3 weeks after the end of cycle 2 (each cycle is 14 days)
  MRD-positive status was defined as FCM positivity in two consecutive BM samples at a 2-week interval, PCR positivity in two consecutive BM samples at a 2-week interval, or both FCM and PCR positivity in a single BM sample after the first-month post-HSCT. Positive FCM was defined as >0.01% of cells with a LAIPs phenotype in >1 BM samples after transplantation. The expressions of leukemia-associated genes were evaluated by TaqMan-based RT-PCR, including Wilms' tumor gene 1 (WT1) and genes which were determined in the diagnostic specimens.
objective remission rate（ORR） | 2 to 3 weeks after the end of cycle 1 (each cycle is 14 days)
  The percentage of people in a study or treatment group who have a partial response or complete response to the treatment within a certain period of time.
objective remission rate（ORR） | 2 to 3 weeks after the end of cycle 2 (each cycle is 14 days)
  The percentage of people in a study or treatment group who have a partial response or complete response to the treatment within a certain period of time.
Progression-free survival (PFS) | Throughout the whole research process, assessed up to 24 months
  From date of Ven plus CAG therapy beginning until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Overall survival | Throughout the whole research process, assessed up to 24 months
  From date of Ven plus CAG therapy beginning until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
The incidence of adverse events | Throughout the whole research process, assessed up to 24 months
  According to Common Terminology Criteria for Adverse Events, CTCAE, V5.0, assessed up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jing Yu, M.D., Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Undecided